CLINICAL TRIAL: NCT07385755
Title: Efficacy of Desvenlafaxine in the Preventive Treatment of Frequent Migraines -- Multicenter, Prospective, Randomized, Controlled Study
Brief Title: Desvenlafaxine for Preventive Treatment of Frequent Migraines
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wensheng Qu, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20251111migraine
Record Dates: First submitted 2026-01-13; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desvenlafaxine (Experimental)
  Interventions: Drug: Desvenlafaxine
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desvenlafaxine — Desvenlafaxine
  Arms: Desvenlafaxine
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
To evaluate whether Desvenlafaxine can reduce the frequency and severity of migraine attacks in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants must be males or females aged 18 years or older
2. Headache meets the diagnostic criteria for episodic migraine according to ICHD-3; with at least a one-year history of migraines and onset before age 50. During the three months prior to the screening visit (one month defined as four weeks), participants must have experienced≥4 and <15 episodes of moderate to severe headaches per month, and had at least ≥6 migraine days within a 4-week run-in period.
3. Obtain the patient's informed consent.

Exclusion Criteria:

1. Have a history of allergy to Desvenlafaxine, or have used Desvenlafaxine within 4 weeks prior to the start of the treatment period
2. Are currently taking or require concomitant administration of contraindicated medications as stated in the package insert, such as monoamine oxidase inhibitors (MAOIs).
3. Comorbid with other types of headaches, such as trigeminal autonomic cephalalgias, more than one episode of tension-type headache per month, or secondary headaches (e.g., those caused by intracranial infections, craniocerebral trauma, cerebrovascular diseases)
4. Severe psychiatric disorders, such as schizophrenia; poorly controlled epilepsy, cognitive impairments, and other chronic pain conditions; serious concomitant medical illnesses that pose significant health risks, including uncontrolled hypertension, cardiac disease, hepatic dysfunction, renal insufficiency, infections; any medical condition or prior surgery likely to affect the absorption, metabolism, or excretion of the study medication
5. Use of venlafaxine analogues, such as serotonin-norepinephrine reuptake inhibitors (SNRIs); unstable use of other types of preventive medications for migraine, including calcitonin gene-related peptide (CGRP) antagonists, topiramate, etc. (≥3 months)
6. Meet the diagnostic criteria for chronic migraine and medication overuse (MO); alcohol dependence or substance use
7. Inability to comprehend the study protocol due to factors including but not limited to low educational attainment, impaired verbal/language function, visual or auditory deficits; failure to accurately complete research documentation (e.g., headache diaries) or incapacity to engage with assessment instruments
8. Female subjects who are trying to conceive, pregnant or breastfeeding, and those not using contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
the change from baseline in monthly migraine days during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12) | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  the change from baseline in monthly migraine days during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)

SECONDARY OUTCOMES:
Days with migraine every 4 weeks during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12) | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Days with migraine every 4 weeks during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
Moderate/severe headache days during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12) | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Moderate/severe headache days during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
The rate of effective responders during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12) | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Treatment effectiveness criterion: reduction in headache days by ≥50% during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
Headache severity during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12) | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  The VAS score reflects the severity of headache pain during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
Cumulative headache duration during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12) | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Based on the headache diary recordings, the cumulative duration of headache episodes will be summed to calculate the total headache time during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
Change in Anxiety and Depression Scores | during the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  Change from baseline in anxiety and depression levels, assessed by the Hospital Anxiety and Depression Scale (HADS). Total score ranges from 0 to 21 for anxiety and 0 to 21 for depression subscales, where 0-7 = normal, 8-10 = borderline, 11-21 = abnormal. Higher scores indicate worse anxiety/depression.
Changes in daily life behavioral capabilities | During the 12-week intervention period (reported in 4-week intervals: Weeks 0-4, 5-8, and 9-12)
  The HIT-6 questionnaire measures the adverse impact of headache on daily functioning in six domains (pain, social functioning, role functioning, vitality, cognitive functioning, psychological distress).

CONTACTS AND LOCATIONS:
Overall Officials: Wensheng Qu, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
No immediate plans exist for IPD sharing, but controlled access may be considered post-study completion